CLINICAL TRIAL: NCT02726919
Title: Prospective Open Label Evaluation of Clobazam Adjunctive Treatment of Adults With Refractory Focal Epilepsy: A Pilot Study
Brief Title: Clobazam Adjunctive Treatment of Adults With Refractory Focal Epilepsy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Pavel Klein (Other)
Collaborators: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor-Investigator, Pavel Klein, Director, Mid-Atlantic Epilepsy and Sleep Center, LLC
Organization: Mid-Atlantic Epilepsy and Sleep Center, LLC (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: maes 007
Record Dates: First submitted 2015-03-13; First posted 2016-04-04 (Estimated); Last update posted 2017-03-23 (Actual); Status verified 2016-03

CONDITIONS: Epilepsy
Keywords: focal epilepsy; clobazam
MeSH Terms: conditions — Epilepsy; Epilepsies, Partial | interventions — Clobazam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Clobazam treatment (Other): This will be an open label study comparing seizure frequency during 12 weeks of baseline observation period with seizure frequency during 16 weeks of clobazam adjunctive treatment
  Interventions: Drug: Clobazam

INTERVENTIONS:
Drug: Clobazam — Following a baseline of 12 weeks patients will be started on clobazam, administered orally in b.i.d. schedule. In patients in whom seizure diaries have been kept prospectively prior to study screening visit, retrospective baseline will be accepted. Patients will be titrated up to either seizure freedom, to side effects or to 40 mg/day, whichever comes first
  Other Names: Onfi

SUMMARY:
The goal of the present study is to obtain pilot data on efficacy and safety of clobazam add-on treatment on adults with drug-resistant focal epilepsy.

This will be an open label study comparing seizure frequency during 12 weeks of baseline observation period with seizure frequency during 16 weeks of clobazam adjunctive treatment. 10 adults aged 18-65 with focal seizures that have failed to respond to ≥ 4 antiepileptic drugs (AEDs) +/- respective surgery will be enrolled. Following a baseline of 12 weeks patients will be started on clobazam, administered orally in b.i.d. schedule. In patients in whom seizure diaries have been kept prospectively prior to study screening visit, retrospective baseline will be accepted. Patients will be titrated up to either seizure freedom, to side effects or to 40 mg/day, whichever comes first. Titration rate will be not be forced. It is anticipated that the majority of subjects will have a 4 week-long titration period. After maximum dose is achieved, maintenance treatment will last for 12 weeks.

DETAILED DESCRIPTION:
Approximately 35 % of patients with epilepsy do not respond to treatment with medications. There is a need for new treatment of refractory focal epilepsy. Clobazam was approved in 2011 in the US for treatment of refractory seizures in patients with Lennox Gastaut syndrome (LGS). Patients with LGS have different seizure types. While pivotal studies evaluated primary generalized seizures, LGS patients also have focal seizures. The goal of the present study is to obtain pilot data on efficacy and safety of clobazam add-on treatment on adults with drug-resistant focal epilepsy.

This will be an open label study comparing seizure frequency during 12 weeks of baseline observation period with seizure frequency during 16 weeks of clobazam adjunctive treatment. 10 adults aged 18-65 with focal seizures that have failed to respond to ≥ 4 antiepileptic drugs (AEDs) +/- respective surgery will be enrolled. Following a baseline of 12 weeks, patients will be started on clobazam, administered orally in b.i.d. schedule. In patients in whom seizure diaries have been kept prospectively prior to study screening visit, retrospective baseline will be accepted. Patients will be titrated up to either seizure freedom, to side effects or to 40 mg/day, whichever comes first. Titration rate will be not be forced. It is anticipated that the majority of subjects will have a 4 week-long titration period. After maximum dose is achieved, maintenance treatment will last for 12 weeks.

Primary efficacy outcome measure will be seizure freedom for 3 months of maintenance treatment with the highest tolerated clobazam dose. Secondary outcome measures will include >75% seizure frequency reduction and median seizure frequency reduction for the whole treatment duration and for the maintenance treatment period, comparing seizure frequency per 28 day periods during treatment vs. baseline. Primary safety outcome measures will include treatment emergent adverse events, and treatment discontinuation due to treatment emergent adverse events.

The number of subjects will be small, n=10. It is therefore likely that results obtained in the present study will not be statistically significant. The goal of the present study is to ascertain whether clobazam add-on treatment in adults with refractory focal epilepsy gives a signal of efficacy greater than that demonstrated with other second and third generation anticonvulsants such as levetiracetam, pregabalin, lacosamide and perampanel; specifically whether clobazam adjunctive treatment shows a trend towards 75% response and seizure freedom rate that surpasses those seen in phase 3 levetiracetam, pregabalin, lacosamide and perampanel studies. The results, if positive, will be used to design a larger controlled study would follow.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-65
2. Stable focal epilepsy, with partial complex seizures including partial complex seizures with or without secondary generalization, partial simple seizures with a clear motor component with or without secondary generalization, and partial simple seizures with secondary generalization.
3. Stable AED doses for at least 30 days
4. Epilepsy duration for > 2 years
5. Past/current treatment with > 4 AEDs. Vagal nerve stimulator treatment will be allowed and will not count as an AED. VNS setting must be stable for 3 months prior to enrollment.
6. Seizure frequency of ≥1/month

Exclusion Criteria:

1. Primary generalized epilepsy
2. Simple partial seizures without motor components or secondary generalization
3. Non-epileptic seizures
4. Progressive neurological disease including neoplasm, CNS degenerative disorders including Alzheimer's disease, other forms of dementia
5. Any systemic illness or unstable medical condition that might pose additional risk, including renal or liver disease, clinically uncontrolled cardiac disease, other unstable metabolic or endocrine disturbances, and active systemic cancer
6. Change in the dose of any Antiepileptic Drug within 30 days prior to enrollment
7. Psychosis within six months of enrollment.
8. Active drug or alcohol dependence or any other factors that, in the opinion of the site investigators would interfere with adherence to study requirements;
9. Pregnancy
10. Use of any CNS-active investigational drugs within 3 months of enrollment.
11. Inability or unwillingness of subject or legal guardian/representative to give written informed consent.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2015-02; Primary Completion 2018-06 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
seizure freedom | 12 weeks
  seizure freedom for 3 months of maintenance treatment with the highest tolerated clobazam dose

SECONDARY OUTCOMES:
>75% seizure frequency reduction and median seizure frequency reduction for the whole treatment duration | 16 weeks
  Secondary outcome measures will include >75% seizure frequency reduction and median seizure frequency reduction for the whole treatment duration and for the maintenance treatment period, comparing seizure frequency per 28 day periods during treatment vs. baseline.
median seizure frequency reduction for the whole treatment duration | 16 weeks
  median seizure frequency reduction for the whole treatment duration
comparing seizure frequency per 28 day periods during treatment vs. baseline | 16 weeks
  comparing seizure frequency per 28 day periods during treatment vs. baseline
quality of life questionnaire (QOLIE-31-P) scores | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Pavel Klein, M.D., Principal Investigator — Mid-Atlantic Epilepsy and Sleep Center
Locations (1):
- MidAtlantic Epilepsy and Sleep Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided